CLINICAL TRIAL: NCT06754774
Title: Shoulder Endurance Test : Valeurs Normatives Chez Une Population De Handballeuses De 14 À 18 Ans En Structures Intensives D'entrainement. SET-HANDBALL
Brief Title: Shoulder Endurance Test: Normative Values in a Population of Female Handball Players Aged 14 to 18 in Intensive Training Structures.
Acronym: SET-HANDBALL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC23.0027
Record Dates: First submitted 2024-08-30; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Healthy Subjects 14 to 18 Years Old
Keywords: Shoulder Endurance Test

STUDY DESIGN:
Intervention Model Description: shoulder endurance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All subjects will perform the same tests.
  Interventions: Diagnostic Test: Shoulder Endurance Test

INTERVENTIONS:
Diagnostic Test: Shoulder Endurance Test — Each patient receive the same intervention, the Shoulder Endurance Test (SET). The Shoulder Endurance Test assesses the endurance of the shoulder muscles in an open kinetic chain.

SUMMARY:
57% of young female handball players experience shoulder pain. This pain is likely to affect training and performance, but most players continue to play despite it. Endurance of the shoulder lateral rotators is a risk factor for sports such as handball. A protocol for applying the Shoulder Endurance Test (SET) to assess the endurance of the lateral rotators of the shoulder has been proposed, but the authors stress the need for further research to validate this test in different sports and for different populations.

The purpose of the study was to determine normative values for the Shoulder Endurance Test in female handball players aged 14 to 18 in intensive training facilities.

ELIGIBILITY:
Inclusion Criteria:

Girls aged 14 to 18 playing handball Handballers training at the Pôle Espoirs or the Centre Labellisé d'Entrainement 29 Players of legal age who have given their consent Signature of consent by parents for underage players

Exclusion Criteria:

Refusal of the minor to take part, even if the legal representatives want the player to take part in the study Refusal to perform the test

Pain preventing the test from being performed

All musculoskeletal conditions affecting the upper limb less than 6 months old.

Shoulder and cervical spine surgery less than 6 months old.

All musculoskeletal conditions affecting the cervical spine less than 6 months old.

Player under legal protection (guardianship/trusteeship) or deprived of liberty

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
To determine normative values for the Shoulder Endurance Test in female handball players aged 14 to 18. | Day 1

SECONDARY OUTCOMES:
Assessing intra-examiner reliability | two months after the test
  Evaluate intra-examiner reliability: on site SET score versus SET score on video analysis (carried out 2 months after the face-to-face test).
Assessing inter-examiner reliability | two months after the test
  Evaluate inter-examiner reliability: SET score for operator 1 versus operator 2 based on analysis of videos
Determine the SET score on the non-dominant arm | Day 1
Evaluate the effort perceived during the test | Day 1
  Borg scale after SET

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided